CLINICAL TRIAL: NCT01428102
Title: Validation of the RapidTEG™ MA Compared to Kaolin in Trauma and Cardiac Patients.
Brief Title: RapidTEG MA Validation
Acronym: R-TEG MA
Status: Terminated | Type: Observational
Why Stopped: Terminiated for trial redesign
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100267A
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Coagulation; Platelet Function
Keywords: Thromboelastography; TEG; Coagulation; RapidTEG; Kaolin
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RapidTEG: Samples tested with TEG which are both citrated and non-citrated and are activated using the reagent RapidTEG.
- Kaolin: Samples tested with TEG which are both citrated and non-citrated and are activated using the reagent Kaolin.

SUMMARY:
During normal physiological conditions hemostasis (the ability of blood to clot) is kept in homeostatic balance by feedback mechanisms. These mechanisms involve an extremely complex series of steps on both sides of the coagulation cascade including cellular components (i.e. clot formation and breakdown). However, should this homeostatic balance be upset, normal hemostasis is affected resulting in pathological clotting (vessel blockage) or bleeding (hemorrhage). In instances that include acquired or congenital abnormalities of the hemostatic system it is clinically important to diagnose, monitor and manage the patient to optimize therapeutic intervention. Moreover, it is important to regulate the hemostasis system in the post-surgical outpatient who receives oral anticoagulant therapy to maintain the homeostatic balance.

The TEG® analyzer, using a small whole blood sample, documents the interaction of platelets with the protein coagulation cascade from the time of placing the blood in the analyzer until initial fibrin formation, clot rate strengthening and fibrin-platelet bonding via GPIIb/IIIa, through eventual clot lysis. It displays both qualitatively and quantitatively the two distinct parts of hemostasis - the part that produces the clot and the part that causes the breakdown of the clot. It shows the balance or degree of imbalance in the patient's hemostasis system, highlights any areas of deficiency or excess, and offers a precise view of the patient's hemostasis condition. If the system is not in balance, one can see where the imbalance lies. If a patient is bleeding, it is crucial to determine the cause of bleeding as soon as possible in order to start the proper treatment.

By utilizing a kaolin/tissue factor activator (RapidTEG™), the TEG® system can measure the interaction and simultaneous contribution of the intrinsic and extrinsic coagulation pathways which initiate and result in clot formation. This RapidTEG™ reagent can deliver results faster than activating with Kaolin alone. This protocol will specifically assess one algorithm called MA. MA is a direct function of the maximum dynamic properties of fibrin and platelet bonding via GPIIb/IIIa that represents the ultimate strength of the fibrin clot. This represents platelet function.

The objective of the study is to demonstrate the substantial equivalence of MA RapidTEG vs. MA Kaolin.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old
* Patient is either a Trauma patient OR is diagnosed with known cardiovascular disease.
* Samples must be tested within the recommended timeline (4-6 minutes for non-citrated and between 15 minutes and 2 hours for citrated)

Exclusion Criteria:

* Patients who have been placed on anticoagulation prophylaxis for other conditions (not CPB/PCI related).
* Patients who have established hemostasis system abnormalities (congenital or other).
* Samples identified as affected by testing errors by lab staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient is either a Trauma patient OR is diagnosed with known cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Correelation of Kaolin to RapidTEG | Concurrent sample tested <2hrs from blood draw
  TEG paramaters were to be correlated in samples run concurrently using Kaolin and RapidTEG assays.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sinai Center for Thrombosis Research, Baltimore, Maryland
  - Univserity of Tennessee Health Sciences Center, Knoxville, Tennessee